CLINICAL TRIAL: NCT02426307
Title: Subclinical Aortic Valve biOprosthesis thRombosis Assessed With 4D Computed tomographY Imaging
Brief Title: Subclinical Aortic Valve Bioprosthesis Thrombosis Assessed With 4D CT
Acronym: SAVORY
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, Associated Professor, Rigshospitalet, Denmark
Other Study IDs: RIGHS.HJE.01
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Thrombosis; Cardiovascular disease; Oral anticoagulation; bioprosthesis; Multidetector Computed Tomography
MeSH Terms: conditions — Aortic Valve Stenosis; Thrombosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transcatheter Aortic Valve Replacement: TAVR: Portico (St Jude Medical), CoreValve (Medtronic), Lotus (Boston Scientific), Edwards Sapien 3 (Edwards LifeSciences),
  Interventions: Procedure: TAVR
- Surgical aortic valve replacement: SAVR: Perimount (Edwards), Epic (St Jude Medical), Trifecta (St Jude Medical)
  Interventions: Procedure: SAVR

INTERVENTIONS:
Procedure: TAVR — TAVR: Transcatheter Aortic Valve Replacement
  Groups: Transcatheter Aortic Valve Replacement
Procedure: SAVR — SAVR: surgical Aortic Valve Replacement
  Groups: Surgical aortic valve replacement

SUMMARY:
TAVR is an increasingly used technique for the treatment of aortic valve stenosis. However, recent clinical experience has suggested that subclinical aortic valve bioprosthesis thrombosis may occur early after valve replacement. The frequency of this potentially ominous phenomenon on both transcatheter and surgical aortic valve bioprosthesis is unknown, as this condition is difficult to detect.

The recent development of cardiac 4D computed tomography imaging (4DCT) shows great promise for the evaluation of valve leaflet mobility and morphology.

The purpose of this study is in an observational design to assess the frequency of subclinical abnormal leaflet motion and morphology in patients treated with transcatheter or surgical aortic valve bioprosthesis. In addition, the 'natural evolution' of this phenomenon as well as its relation to medical treatment and MACCE will be assessed.

DETAILED DESCRIPTION:
MATERIAL In the period from May 2014 to November 2015, a random subset of patients who underwent transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR) were offered intensified post-procedural clinical and imaging follow-up. It is intended to examine a variety of implanted transcatheter heart valves (THV) as well as surgical aortic valve bioprosthesis.

METHODS:

Post-procedural clinical and imaging follow-up encompasses the following:

* Thoracic 4DCT scanning - with evaluation of leaflet morphology and leaflet motion
* Transthoracic echocardiography - with evaluation of peak aortic valve gradient, mean aortic valve gradient, aortic valve area/effective orifice area (cm2), paravalvular leakage, central aortic valve regurgitation, and left ventricular ejection fraction
* Clinical follow-up: improvement in New York Heart Association (NYHA) class dyspnea, and major adverse cardiac and cerebro-vascular events (MACCE)
* Registration of anti-coagulation/anti-thrombotic therapy following aortic valve replacement

All patients will receive the above-described post-procedural follow-up at two different time-points:

* The first follow-up contact will be planned 30 to 180 days after the TAVR or SAVR procedure. The medical treatment will not be changed based on the generated data.
* The second follow-up contact will be planned 120 to 180 days after the first follow-up contact (see above). This second follow-up offers the possibility to study the 'natural evolution' of this process. In those patients with an abnormal leaflet morphology and/or motion, a treatment with rivaroxaban 20mg daily will be initiated.
* Those patients initiated on rivaroxaban after the second follow-up will be called in for a third clinical and imaging follow-up, with focus on leaflet morphology and/or motion after rivaroxaban therapy. In case of persistent abnormal leaflet morphology and/or motion despite NOAC, a treatment with Marevan (INR 2-3) will be initiated.
* Those patients initiated on Marevan after the third follow-up will be called in for a fourth clinical and imaging follow-up contact.

ELIGIBILITY:
Inclusion Criteria:

Successful TAVR or SAVR performed at Rigshospitalet, Copenhagen, Denmark

Exclusion Criteria:

* renal dysfunction (eGFR <25 ml/min)
* TAVR-in-TAVR
* Patients living in Greenland or the Faroe Islands

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A random subset of patients undergoing transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR) because of aortic valve stenosis.
Sampling Method: Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-09 (Actual); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with abnormal aortic valve bioprosthesis leaflet mobility and morphology | At least 21 days post-procedure

SECONDARY OUTCOMES:
Frequency of abnormal aortic valve bioprosthesis leaflet mobility and morphology | At least 21 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lars Søndergaard, MD, Study Director — Department of Cardiology, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Denmark
Locations (1):
- Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Thyregod HG, Steinbruchel DA, Ihlemann N, Nissen H, Kjeldsen BJ, Petursson P, Chang Y, Franzen OW, Engstrom T, Clemmensen P, Hansen PB, Andersen LW, Olsen PS, Sondergaard L. Transcatheter Versus Surgical Aortic Valve Replacement in Patients With Severe Aortic Valve Stenosis: 1-Year Results From the All-Comers NOTION Randomized Clinical Trial. J Am Coll Cardiol. 2015 May 26;65(20):2184-94. doi: 10.1016/j.jacc.2015.03.014. Epub 2015 Mar 15. PMID 25787196
- [Result] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Derived] Sondergaard L, De Backer O, Kofoed KF, Jilaihawi H, Fuchs A, Chakravarty T, Kashif M, Kazuno Y, Kawamori H, Maeno Y, Bieliauskas G, Guo H, Stone GW, Makkar R. Natural history of subclinical leaflet thrombosis affecting motion in bioprosthetic aortic valves. Eur Heart J. 2017 Jul 21;38(28):2201-2207. doi: 10.1093/eurheartj/ehx369. PMID 28838044